CLINICAL TRIAL: NCT02511522
Title: Phase III Study of Palliative Radiotherapy for Symptomatic Hepatocellular Carcinoma and Liver Metastases
Brief Title: Study of Palliative Radiotherapy for Symptomatic Hepatocellular Carcinoma and Liver Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HE1
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma; Liver Metastases
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Supportive Care (Active Comparator): Patients will be randomized 1:1 to receive best supportive care alone
  Interventions: Other: Best Supportive Care
- Best Supportive Care + RT 8 Gy/1 (Experimental): Patients will be randomized 1:1 to receive best supportive care plus radiation therapy (8 Gy in 1 fraction),
  Interventions: Other: Best Supportive Care; Radiation: Palliative Radiation Therapy

INTERVENTIONS:
Other: Best Supportive Care — Including analgesics, palliative care and/or pain specialist assessment as needed
Radiation: Palliative Radiation Therapy — 8 Gy in 1 fraction in whole liver or near whole liver. Including anti-emetic pre-medications
  Arms: Best Supportive Care + RT 8 Gy/1

SUMMARY:
The purpose of this study is to see whether one dose of palliative radiation therapy directed to the liver in combination with standard BSC might help to reduce liver pain/discomfort due to cancer when compared to getting standard BSC alone.

DETAILED DESCRIPTION:
The standard treatment for liver cancer pain or discomfort like yours is known as best supportive care (BSC) and includes pain-relieving medicines called analgesics. This type of treatment can help in some cases; however, some analgesics require a healthy liver to work properly. This means that there are many patients who have a hard time managing their liver cancer pain/discomfort with BSC alone.

Sometimes radiation therapy is given in the "palliative" setting meaning it is designed to treat the pain/discomfort and not necessarily to shrink or eliminate the tumour. Palliative radiation therapy is often given when patients have painful bone tumours, but is not yet widely used to treat liver pain/discomfort. Palliative radiation therapy is usually given in smaller amounts and less frequently than other kinds of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cancer by at least one criterion listed below:

  * Pathologically or cytologically proven carcinoma from primary site or site of metastases;
  * Pathologically or cytologically proven HCC;
  * HCC diagnosed by standard imaging criteria: arterial enhancement and delayed washout on multiphasic computerized tomography (CT) or magnetic resonance imaging (MRI) in the setting of cirrhosis or chronic hepatitis B or C without cirrhosis.
* Largest burden of cancer in the liver is confirmed with CT scan or MRI corresponding to the clinically painful area done within 120 days prior to randomization.
* Diffuse (infiltrative involving > 50% of the liver), multifocal (> 10 lesions) or locally advanced cancer (at least one lesion > 10cm, vascular invasion, or multiple lesions with at least one > 6cm) involving the liver.
* In the investigator's opinion, patient is unsuitable for or refractory to standard local and regional therapies. For example:

  * HCC unsuitable for resection, radiofrequency ablation (RFA), transarterial chemo embolization (TACE) or radical intent, ablative dose stereotactic body radiation therapy (SBRT);
  * Colorectal carcinoma metastases unsuitable for resection, RFA or radical intent, ablative dose SBRT (e.g. SBRT, > 30 Gy in 5 fractions, may be an option for up to 3 metastases < 5cm each, or up to 5 metastases < 3 cm each).
* Unsuitable for, high risk for, or refractory to, standard systemic chemotherapy or targeted therapy (e.g. sorafenib).
* Patient reports moderate or severe pain/discomfort prior to the baseline evaluation and this pain is considered "stable" over a period of up to 7 days prior to randomization.

Definition of moderate pain:

Patient reports level of 4-6 (on a BPI scale from 0 to 10) pain or discomfort "at its worst in the past 24 hours", occurring in the right upper quadrant of the abdomen, the upper abdomen and/or referred to the right shoulder, attributable to liver cancer.

Definition of severe pain:

Patient reports level of 7-10 (on a BPI scale from 0 to 10) pain or discomfort "at its worst in the past 24 hours", occurring in the right upper quadrant of the abdomen, the upper abdomen and/or referred to the right shoulder, attributable to liver cancer.

Definition of "stable" pain:

Patient must show moderate or severe "stable" pain by reporting a score of 4 or greater (on 2 separate days within the 7 day period prior to randomization) with the difference of these scores being 0, 1, 2 or 3.

* Patient reports moderate or severe pain (i.e. pain score is 4 or higher). This baseline score must also be stable compared to the most recent pre-baseline pain score with the difference between these scores being 0, 1, 2, or 3.
* Blood work obtained within 14 days prior to randomization as follows:

  * Hemoglobin > 70 g/L;
  * Platelets > 25 x 10^9/L
  * Absolute neutrophil count (ANC) > 1.0 x 10^9/L
  * INR < 3;
  * Bilirubin < 2.5 UNL (except for subjects with Gilbert's Disease who are eligible despite elevated serum bilirubin level)
  * AST or ALT < 10 x ULN.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3 within 14 days of Randomization (see Appendix II).
* Life expectancy of > 3 months.
* 18 years of age or older at the time of randomization.
* Patient is willing to complete the Pre-Baseline Pain/Discomfort Questionnaire and the Pain/Discomfort and Medication Questionnaire in English, French or other validated language (please contact the HE.1 Study Coordinator). The baseline assessment must be completed within required timelines prior to randomization. Unwillingness to complete the Pre-Baseline Pain/Discomfort Questionnaire and Pain/Discomfort and Medication Questionnaire will make the patient ineligible for the study.
* Patient is able (i.e. sufficiently fluent) and willing to complete the QoL questionnaires in English, French or other languages in which the FACT-Hep is available. The baseline assessment must be completed within required timelines prior to randomization.

Inability (illiteracy in languages listed above, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the QoL questionnaires will make the patient ineligible for QoL assessment.

* Patient is not pregnant, planning on becoming pregnant or planning on fathering a child in the next 90 days.

Women/men of childbearing potential must have agreed to use a highly effective contraceptive method. A woman is considered to be of "childbearing potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy/vasectomized partner. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures.

Women of childbearing potential will have a pregnancy test to determine eligibility as part of the Pre-Study Evaluation; this may include an ultrasound to rule-out pregnancy if a false-positive is suspected. For example, when beta-human chorionic gonadotropin is high and partner is vasectomized, it may be associated with tumour production of hCG, as seen with some cancers. Patient will be considered eligible if an ultrasound is negative for pregnancy

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate;
* Patients must be accessible for treatment and follow-up. Investigators must ensure the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient randomization (earlier is preferred).

Exclusion Criteria:

* Prior radiotherapy to the upper abdomen that would result in substantial overlap of the irradiated volume (e.g. > 50% of liver receiving > 24 Gy in 2 Gy equivalent dose);
* Prior selective internal radiotherapy directed to the liver or hepatic arterial yttrium therapy, at any time.
* Cholangitis or acute bacterial infection requiring intravenous antibiotics within 28 days prior to study entry.
* Radiographic evidence of intrabiliary cancer within the common or main branches of the biliary system, < 4 months prior to randomization.
* Child-Pugh score greater than C10 (a score of C10 is allowed).
* Chemotherapy or TACE administered within the past 4 weeks.
* Targeted therapy (e.g. Sorafenib) received within the past 2 weeks.
* Plans for chemotherapy, targeted therapy or TACE in the next 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ann Dawson, Study Chair — Univ. Health Network-Princess Margaret Hospital
Locations (7):
- Canada (7):
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dawson LA, Ringash J, Fairchild A, Stos P, Dennis K, Mahmud A, Stuckless TL, Vincent F, Roberge D, Follwell M, Wong RKW, Jonker DJ, Knox JJ, Zimmermann C, Wong P, Barry AS, Gaudet M, Wong RKS, Purdie TG, Tu D, O'Callaghan CJ. Palliative radiotherapy versus best supportive care in patients with painful hepatic cancer (CCTG HE1): a multicentre, open-label, randomised, controlled, phase 3 study. Lancet Oncol. 2024 Oct;25(10):1337-1346. doi: 10.1016/S1470-2045(24)00438-8. Epub 2024 Sep 5. PMID 39245060

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiotherapy Combined With Best Supportive Care: Patients receive a radiation therapy with the use of 8 Gy in one fraction to the whole (or near-whole) liver together with the best supportive care.
- Best Supportive Care Alone: Patients receive only the best supportive care.
Period: Overall Study
Arm/Group | Radiotherapy Combined With Best Supportive Care | Best Supportive Care Alone
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiotherapy Combined With Best Supportive Care | Best Supportive Care Alone | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Median (Full Range); unit: years] | 66 [41 to 88] | 62 [39 to 89] | 65 [39 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 18 | 19 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 33 | 66
ECOG (Eastern Cooperative Oncology Group) Perfromance Status [Count of Participants; unit: Participants] — 0: Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0 | 1 | 0 | 1
    1 | 18 | 8 | 26
    2 | 7 | 13 | 20
    3 | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Significant Improvement of Liver Cancer Pain/Discomfort
Description: • Proportion of patients achieving improvement of liver cancer pain/discomfort by ≥ 2 points in pain "intensity at worst " on Brief Pain Inventory (BPI) from baseline to day 30.
Time Frame: 30 days
Population: All patients who completed both baseline and day 30 assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy Combined With Best Supportive Care | Best Supportive Care Alone
Number analyzed (Participants) | 24 | 18
Participants | 16 | 4
Statistical Analysis 1: Comparison: Radiotherapy Combined With Best Supportive Care vs Best Supportive Care Alone; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Adjusting for stratification factor (Hepatocellular carcinoma versus liver metastases)

2. Secondary Outcome: Proportion of Patients Alive at Day 90.
Description: Estimated by Kaplan-Meier method for overall survival defined as time from randomization to death from any cause.
Time Frame: 90 days
Population: All patients randomized
Measure: Number (95% Confidence Interval); unit: percentage of alive at 90 days
Arm/Group | Radiotherapy Combined With Best Supportive Care | Best Supportive Care Alone
Number analyzed (Participants) | 33 | 33
percentage of alive at 90 days | 51.18 [33.12 to 66.63] | 32.99 [17.46 to 49.42]
Statistical Analysis 1: Comparison: Radiotherapy Combined With Best Supportive Care vs Best Supportive Care Alone; Test type: Superiority; p = 0.068, Log Rank; Stratified Log Rank test adjusting for the stratification factor (Hepatocellular carcinoma versus liver metastases)

3. Secondary Outcome: Proportion of Patients Achieving a 25% Reduction in Opioid Use at 30 Days (Employing Daily Morphine Equivalence Scale).
Time Frame: 30 days
Population: Patients who reported taking opioid medications in the 24 hours prior to their both baseline and day 30 assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy Combined With Best Supportive Care | Best Supportive Care Alone
Number analyzed (Participants) | 14 | 14
Participants | 5 | 3
Statistical Analysis 1: Comparison: Radiotherapy Combined With Best Supportive Care vs Best Supportive Care Alone; Test type: Superiority; p = 0.45, Cochran-Mantel-Haenszel; adjusting for the stratification factor (Hepatocellular carcinoma versus liver metastases)

4. Secondary Outcome: Proportion of Patients Achieving Improvement of Liver Cancer Pain/Discomfort by ≥ 2 Points in Pain "Intensity at Worst " AND With no Increase in Opioid Use (Employing Daily Morphine Equivalence Scale) on BPI From Baseline to 30 Days.
Time Frame: 30 days
Population: Patients who completed both baseline and day 30 pain/discomfort assessments and reported taking opioid medications in the 24 hours prior to their both baseline and day 30 assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy Combined With Best Supportive Care | Best Supportive Care Alone
Number analyzed (Participants) | 14 | 14
Participants | 3 | 0
Statistical Analysis 1: Comparison: Radiotherapy Combined With Best Supportive Care vs Best Supportive Care Alone; Test type: Superiority; p = 0.07, Cochran-Mantel-Haenszel; adjusting for the stratification factor (Hepatocellular carcinoma versus liver metastases)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Only grade 2 or higher adverse events were collected.
Arm/Group | Radiotherapy Combined With Best Supportive Care | Best Supportive Care Alone
All-Cause Mortality (participants affected / at risk) | 19/33 | 24/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 19/33 | 11/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy Combined With Best Supportive Care (N=33) | Best Supportive Care Alone (N=33)
Abdominal pain (Gastrointestinal disorders) | 11 | 5
Constipation (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Fatigue (General disorders) | 5 | 6
Pain (General disorders) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT02511522/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT02511522/SAP_001.pdf